CLINICAL TRIAL: NCT05531357
Title: Physiologic Mechanisms Underlying Ovarian Follicular Waves During the Menstrual Cycle
Status: Completed | Type: Observational
Sponsor: University of Saskatchewan (Other)
Collaborators: Ansh Labs (Unknown)
Responsible Party: Principal Investigator, Angela Baerwald, Associate Professor, University of Saskatchewan
Other Study IDs: Bio 2080
Record Dates: First submitted 2022-08-29; First posted 2022-09-07 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Reproductive Issues
Keywords: ovarian follicles; ovulation
MeSH Terms: interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dried blood spots, serum frozen at -80 C and dried urine spot samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transvaginal ultrasound scans — Transvaginal ultrasound scans to map ovarian follicle growth and ovulation, finger-prick blood sampling for dried blood spot (DBS) hormonal assays and urine sampling for hormone metabolites, every consecutive day for an interovulatory interval.
  Weekly venipuncture samples will be taken for standard ELISA hormonal assays. The hormones of interest are FSH, LH, estradiol, progesterone, AMH, inhibins A and B, GDF-9 and BMP-15.
  Other Names: Finger-prick blood sampling for dried blood spots; Urine sampling; Venipunctures

SUMMARY:
The research aims to characterize changes in ovarian and pituitary hormones associated with the development of ovarian follicular waves during the human menstrual cycle.

DETAILED DESCRIPTION:
Our laboratory's previous research has demonstrated that multiple waves of ovarian follicles develop throughout the menstrual cycle. Approximately 2/3 of women develop 2 follicle waves throughout their cycle while the remainder exhibit 3 waves of follicle growth (1,2). This study is to follow up on those findings to determine how pituitary and ovarian hormones regulate the development of follicle waves in women, with a combination of ultrasound scans and blood and urine sampling to characterize how follicles grow during the menstrual cycle in 50 women of reproductive age. Changes in follicle growth across the cycle will be compared with changes in hormone production.

The new findings will be essential for improving understanding of female reproduction, with clinical applications in contraception, fertility and menopausal care for women across their reproductive lifespan.

ELIGIBILITY:
Inclusion Criteria:

* Healthy biological females
* Regular menstrual cycles (21-35 days)

Exclusion Criteria:

* BMI <18 or >30
* Pregnancy
* Breastfeeding mothers
* Current infertility
* History of hysterectomy or oophorectomy
* Reproductive health issues that can interfere with study outcomes
* Smoking
* Metabolic syndrome (blood pressure, fasting glucose, fasting insulin and serum lipids measured to assess eligibility)
* Not on any hormonal medication that affects reproduction (including hormonal contraception)
* Hyperprolactinemia
* Abnormal thyroid stimulating hormone assay

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers who respond to advertisements placed in the community, local offices and the University of Saskatchewan's website
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-09-17 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Antral follicle diameter | One menstrual cycle (21-35 days) per volunteer
  Daily diameters of individual follicles ≥ 2mm from ultrasound examination
Antral follicle count | One menstrual cycle (21-35 days) per volunteer
  Daily count of the number of follicles >2 mm from ultrasound examination
Follicle stimulating hormone (FSH) serum level | One menstrual cycle (21-35 days) per volunteer
  Daily measurements of FSH in IU/L
Luteinizing hormone (LH) serum level | One menstrual cycle (21-35 days) per volunteer
  Daily measurements of LH in IU/L
Estradiol serum level | One menstrual cycle (21-35 days) per volunteer
  Daily measurements of estradiol in pg/mL
Progesterone serum level | One menstrual cycle (21-35 days) per volunteer
  Daily measurements of progesterone in ng/mL
Anti-mullerian hormone (AMH) serum level | One menstrual cycle (21-35 days) per volunteer
  Daily measurements of AMH in ng/mL
Inhibin A serum level | One menstrual cycle (21-35 days) per volunteer
  Daily measurements of inhibin A in pg/mL
Inhibin B serum level | One menstrual cycle (21-35 days) per volunteer
  Daily measurements of inhibin B in pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Angela R Baerwald, PhD,MD,CCFP, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baerwald AR, Adams GP, Pierson RA. A new model for ovarian follicular development during the human menstrual cycle. Fertil Steril. 2003 Jul;80(1):116-22. doi: 10.1016/s0015-0282(03)00544-2. PMID 12849812
- [Background] Baerwald AR, Adams GP, Pierson RA. Characterization of ovarian follicular wave dynamics in women. Biol Reprod. 2003 Sep;69(3):1023-31. doi: 10.1095/biolreprod.103.017772. Epub 2003 May 14. PMID 12748128